CLINICAL TRIAL: NCT04419519
Title: Veneto-STOP Study: Sequential Assessment of Minimal Residual Disease by Next Generation Sequencing to Optimize Outcomes and Minimize Exposure in Venetoclax-Treated CLL/SLL Patients
Brief Title: Assessing Minimal Residual Disease by Next- Generation Sequencing to Minimize Exposure in People With CLL or SLL Who Have Been Treated With Venetoclax
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Adaptive Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-395
Record Dates: First submitted 2020-06-04; First posted 2020-06-05 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL)
Keywords: Venetoclax; Anti-CD20 monoclonal antibody; 19-395
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — venetoclax

STUDY DESIGN:
Intervention Model Description: This is a multicenter clinical stopping trial for venetoclax-treated chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) patients.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Venetoclax monotherapy (Experimental)
  Interventions: Drug: Venetoclax monotherapy
- Venetoclax with anti-CD20 monoclonal antibody (Experimental)
  Interventions: Drug: Venetoclax with anti CD20 monoclonal antibody

INTERVENTIONS:
Drug: Venetoclax monotherapy — Venetoclax monotherapy
  Arms: Venetoclax monotherapy
Drug: Venetoclax with anti CD20 monoclonal antibody — Venetoclax with anti CD20 monoclonal antibody
  Arms: Venetoclax with anti-CD20 monoclonal antibody

SUMMARY:
This study will find out whether people with CLL or SLL who have received treatment with venetoclax, either alone or in combination with another drug, and who are found to be MRD-negative, can stop treatment with venetoclax and remain off-treatment for 12 months or more. The researchers will also see whether study participants remain MRD-negative after they stop treatment with venetoclax.

DETAILED DESCRIPTION:
Screening Phase:

Patients will be identified by clinical investigators at participating centers. Patients who sign the screening consent will undergo MRD assessment with the clonoSEQ® assay. If the assessment identifies the patient to be MRD negative, the patient will undergo a repeat MRD assessment ≥ 28 days later. If two consecutive MRD assessments indicate MRD-negativity, the patient will then sign the study intervention phase informed consent form and will undergo the rest of the screening process.

Enrollment

Once the patient fulfills all eligibility criteria, the patient will be enrolled into one of two cohorts based on the type of therapy they are receiving at the time of enrolled:

Cohort A: Venetoclax monotherapy at time of enrollment.

Cohort B: Venetoclax with anti CD20 monoclonal antibody at time of enrollment (The latter includes patients who initiated anti CD20 monoclonal antibody with venetoclax and have since completed the anti CD20 monoclonal antibody portion of the regimen.)

ELIGIBILITY:
Screening Phase Inclusion Criteria:

* ≥ 18-years-old
* Diagnosis of chronic lymphocytic leukemia or small lymphocytic lymphoma confirmed by the enrolling institution
* Receiving treatment or planning to receive treatment within 30 days with a venetoclax-based regimen as defined below:

  * Venetoclax monotherapy
  * Venetoclax in combination with anti CD20 monoclonal antibody (Patients must have completed the anti CD20 monoclonal antibody portion of the regimen prior to discontinuing therapy)
* Patient has or will have specimen to identify the CLL or SLL clone(s) for future MRD assessments by clonoSEQ® defined as any of the following:

  * 3-5 bone marrow aspirate slides (banked), 3-5 FFPE slides (banked), banked tumor cells or banked DNA collected from the patient at any time from original diagnosis of CLL or SLL to present
  * Peripheral blood, marrow, or lymph node involvement for fresh sample collection
* The screening ID sample (high disease burden sample) can be sent prior to start of venetoclax-based therapy to identify the clone for tracking.

Study Intervention Phase Inclusion Criteria:

* Patients must have received venetoclax-based therapy for at least 6 months (including dose interruptions)
* If receiving venetoclax in combination with anti-CD20 monoclonal antibody, patients must have completed or discontinued the anti CD20 monoclonal antibody portion of the regimen prior to discontinuing therapy
* Patients must have two MRD-negative assessments (defined by ≥ 10^-5 sensitivity) on the peripheral blood by the clonoSEQ® assay at least 28 days apart. Given that MRD status is a dynamic endpoint which may improve with time, if a patient is screen failure based on MRD status (i.e. MRD positive at the 10-5 sensitivity), they may be rescreened to assess for study eligibility.
* Patients must have achieved a complete or partial remission with the venetoclax-based regimen. Criteria for remission are per iwCLL 2018 guidelines. For this protocol, bone marrow biopsy/aspirate evaluation is not necessary to determine remission status.

Exclusion Criteria (both study phases):

* Ongoing participation in a clinical trial that supplies venetoclax and/or anti CD20 monoclonal antibody
* Unwilling or unable to participate in all required study evaluations and procedures.
* Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local patient privacy regulations).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients able to remain off CLL/SLL directed therapy | 2 years
  This will be described as a percentage of all patients with available data at 12 cycles of follow up (evaluable population).

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Thompson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Memorial Sloan Kettering Basking Ridge (All protocol activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (All protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All protocol activities), Harrison, New York
  - Columbia University, New York, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Uniondale, New York
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm